CLINICAL TRIAL: NCT02468973
Title: Accompanying and Supporting Patients in Lifestyle Health Behavior Change by Medical Students at Primary Care Clinics in Zefat Israel
Brief Title: Supporting Patients in Lifestyle Health Behavior Change by Medical Students at Primary Care Clinics in Zefat Israel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Dr Lilach Maletsky, MD, Clalit Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: COM-0046-14
Record Dates: First submitted 2015-05-26; First posted 2015-06-11 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Life Style
Keywords: health behavior; consultation; undergraduate
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Life style counseling (Other): Students will meet chronic patients and will counsel for life style
  Interventions: Behavioral: Life style counseling

INTERVENTIONS:
Behavioral: Life style counseling — Life style counseling for chronic patients by medical students

SUMMARY:
Medical students from zefad medical school volunteer to assist patients with chronic diseases to make lifestyle changes.

Each student will work closely with a family doctor who finds patients who need and want it accompanied by a change he introduced them and guide him on health status, medication and change the desired objectives.

In the program students will receive guidance on healthy lifestyle and support a patient to perform health changes in theoretical and practical. Training sessions will be held periodically, close supervision and guidance, counseling and cross-fertilization and updates from the scientific literature.

DETAILED DESCRIPTION:
The challenge of the third millennium doorway medicine is dealing with an epidemic of chronic diseases caused by unhealthy lifestyle. Medical students spent many hours in acquiring knowledge in the medical professions but little time invested in studying fields related to medicine lifestyles.

On the other side, the family doctors in charge of health promotion in the community find themselves inundated with patients that often can make lifestyle on the one hand but a huge shortage of time for providing advice and support in favor of this issue on the other.

The Faculty of Medicine in Safed project exists "As you hear" where each student is asked to choose a project support and assistance to the community. Medical students who elected to be incorporated into this project with the assistance of patients with chronic diseases to lifestyle changes.

Each student will work closely with a family doctor who finds for patients who need and want it accompanied by a change he introduced them and guide him on health status, medication and change the desired objectives.

In the program students will receive guidance on healthy lifestyle and support a patient to perform health changes in theoretical and practical. Training sessions will be held periodically, close supervision and guidance, counseling and cross-fertilization and updates from the scientific literature.

The student will meet with patients and support them to make a lifestyle change in favor of health

ELIGIBILITY:
Inclusion Criteria:

* aged 20-80
* male or female
* Chronically ill patients who suffers from hypertension, diabetes, obesity, stable heart disease, high blood lipids, etc
* spotted by a family doctor needed a change in lifestyle to improve his health
* expressed his desire to participate process consulting and support.

Exclusion Criteria:

* patients aged less than 20 or more than 80 years
* patients with complex medical problems and unstable heart disease
* patients who are not interested in supporting.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
patients report of lifestyle change | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: lilach malatskey, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Clalit Health Center, Safed, Israel